CLINICAL TRIAL: NCT05764525
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Parallel Group, Placebo-Controlled Study to Evaluate the Efficacy and Safety of VVZ-149 Injections for the Treatment of Postoperative Pain Following Laparoscopic Colectomy
Brief Title: Efficacy and Safety of VVZ-149 Injections in Patients Undergoing Laparoscopic Colectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vivozon Pharmaceutical Inc. (Industry)
Responsible Party: Sponsor
Organization: Vivozon, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VVZ149-POP-P3-K301
Record Dates: First submitted 2023-02-28; First posted 2023-03-10 (Actual); Results first posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Pain, Postoperative; Acute Pain
MeSH Terms: conditions — Pain, Postoperative; Acute Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- VVZ-149 Injections (Experimental)
  Interventions: Drug: VVZ-149 Injections
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VVZ-149 Injections — IV infusion of 1000 mg of VVZ-149
  Other Names: Opiranserin Injections
  Arms: VVZ-149 Injections
Drug: Placebo — IV infusion of 0 mg of VVZ-149
  Arms: Placebo

SUMMARY:
The purpose of this phase 3 study is to evaluate the efficacy and safety of VVZ-149 Injections for the treatment of postoperative pain following laparoscopic colectomy.

ELIGIBILITY:
Inclusion Criteria:

* Men and women who are at least 18 years of age
* Female subjects who are not pregnant or breastfeeding
* Subjects undergoing a planned first laparoscopic colectomy
* Subjects classified in American Society of Anesthesiologists (ASA) risk class of I or II
* Subjects who report the pain intensity ≥ 5 on the NRS measured after surgery
* Subjects who have the ability to understand study procedures and communicate clearly with the investigator and staff
* Subjects who provide written informed consent prior to participation in the study

Key Exclusion Criteria:

* Subjects undergoing emergency or unplanned surgery
* Subjects who had a previous laparoscopic colectomy procedure, or who had any laparoscopic resection procedure
* Subjects with pre-existing conditions causing preoperative pain at the site of surgery
* Female subjects who are pregnant or breastfeeding
* Diagnosis of chronic pain (e.g., persistent pain with the intensity of NRS ≥ 5 at baseline)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2021-07-19 (Actual); Primary Completion 2022-11-03 (Actual); Study Completion 2022-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Doo Lee, PhD, Study Chair — Vivozon Pharmaceutical Inc.
Locations (5):
- South Korea (5):
  - Asan Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Bundang Hospital, Seoul
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Lee HJ, Sim JY, Song I, Nedeljkovic SS, Kim DK, Oh AY, Yoon SZ, Moon YJ, Park MH, Park I, Kim J, Lee SR, Cho S, Bahk JH. Reduction of postoperative pain and opioid consumption by VVZ-149, first-in-class analgesic molecule: A confirmatory phase 3 trial of laparoscopic colectomy. J Clin Anesth. 2025 Feb;101:111729. doi: 10.1016/j.jclinane.2024.111729. Epub 2024 Dec 19. PMID 39705738

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | VVZ-149 Injections | Placebo
Started (Randomized) | 142 | 143
Treated | 141 | 143
Completed | 136 | 135
Not Completed | 6 | 8
Not completed — Inclusion/exclusion criteria not met Inclusion/exclusion criteria not met | 1 | 0
Not completed — Withdrawal by Subject | 4 | 8
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VVZ-149 Injections | Placebo | Total
Number analyzed (Participants) | 141 | 143 | 284
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 91 | 72 | 163
  >=65 years | 50 | 71 | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (9.66) | 62.8 (9.76) | 61.8 (9.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 59 | 121
  Male | 79 | 84 | 163
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 141 | 143 | 284
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  South Korea | 141 | 143 | 284
BMI [Mean (Standard Deviation); unit: kg/m2] | 24.66 (3.044) | 24.21 (2.610) | 24.44 (2.838)

OUTCOME MEASURES:

1. Primary Outcome: Time-weighted Sum of Pain Intensity Differences for 12 Hours Post-dose (SPID 12)
Description: Pain Intensity (PI) was assessed on an 11-point numerical rating scale from 0 (no pain) to 10 (worst pain imaginable). Time-weighted Sum of Pain Intensity Difference (PID) for 12 hours post-dose (SPID 12) was estimated using the linear trapezoidal rule (L x Hour) with the PI scores assigned from Time 0 to Time 12 hours post-dose using the following formula. The theoretical SPID 12 ranges from 0 to 120. A higher value of SPID indicates greater pain relief.
  SPID 12 = S [T(i)-T(i-1)] × [PID(i)+PID(i-1)]/2, when PID(i) =Predose PI-PI at Time i
Time Frame: 0-12 hours post-dose
Population: mITT
Measure: Least Squares Mean (Standard Error); unit: score on a scale*hours
Arm/Group | VVZ-149 Injections | Placebo
Number analyzed (Participants) | 141 | 143
score on a scale*hours | 26.83 (1.73) | 19.89 (1.72)
Statistical Analysis 1: Comparison: VVZ-149 Injections vs Placebo; Test type: Superiority; p = 0.0047, ANOVA; Difference of least squares mean = 6.938, 95% CI 2-sided [2.145 to 11.731]

2. Secondary Outcome: Total Number of Patient-controlled Analgesia (PCA) Requests for 12 Hours Post-dose
Description: Total number of patient-controlled analgesia (PCA) requests from Time 0 to Time 12 hours was compared between the VVZ-149 Injections group and the placebo group.
Time Frame: 0-12 hours post-dose
Population: mITT
Measure: Mean (Standard Deviation); unit: requests
Arm/Group | VVZ-149 Injections | Placebo
Number analyzed (Participants) | 141 | 143
requests
  Time 4-6 Hour | 7.0 (10.24) | 17.6 (63.54)
  Time 6-8 Hour | 5.0 (5.97) | 10.1 (19.79)
  Time 8-10 Hour | 4.6 (6.88) | 8.0 (16.18)

3. Secondary Outcome: Total Amount of PCA and Rescue Medication Consumption for 12 Hours Post-dose
Description: Total amount of PCA and rescue medication consumption from Time 0 to Time 12 hours was compared between the VVZ-149 Injections group and the placebo group.
Time Frame: 0-12 hours post-dose
Population: mITT
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | VVZ-149 Injections | Placebo
Number analyzed (Participants) | 141 | 143
mg
  Time 2-4 Hour | 38.6 (28.28) | 47.0 (32.92)
  Time 4-6 Hour | 24.0 (20.45) | 31.9 (27.00)
  Time 6-8 Hour | 19.1 (19.63) | 27.6 (25.36)
  Time 8-10 Hour | 17.8 (19.64) | 24.9 (24.13)

ADVERSE EVENTS:
Time Frame: 21 days (+7d)
Description: Following laparoscopic colectomy, adverse events were monitored continuously during Time 0 to Time 48 hours and a safety follow-up assessment was performed between Days 21 and 28.
Arm/Group | VVZ-149 Injections | Placebo
All-Cause Mortality (participants affected / at risk) | 0/141 | 0/143
Serious Adverse Events (participants affected / at risk) | 0/141 | 0/143
Other Adverse Events (participants affected / at risk) | 101/141 | 98/143
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | VVZ-149 Injections (N=141) | Placebo (N=143)
Nausea (Gastrointestinal disorders) | 48 | 44
Vomiting (Gastrointestinal disorders) | 19 | 10
Haematochezia (Gastrointestinal disorders) | 10 | 9
Post procedural fever (Injury, poisoning and procedural complications) | 45 | 41
Hypertension (Vascular disorders) | 12 | 11
Phlebitis (Vascular disorders) | 10 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-27): https://cdn.clinicaltrials.gov/large-docs/25/NCT05764525/Prot_SAP_000.pdf